CLINICAL TRIAL: NCT04717986
Title: Dapagliflozin Effects on Mayor Adverse Cardiovascular Events in Patients With Acute Myocardial Infarction (DAPA-AMI). Randomized Clinical Trial
Brief Title: Dapagliflozin Effects on Mayor Adverse Cardiovascular Events in Patients With Acute Myocardial Infarction (DAPA-AMI)
Acronym: DAPA-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Hilda Elizabeth Macías Cervantes, Internist Physician and Master in Clinical Research assigned to the Internal Medicine Service, High Specialty Medical Unit No. 1, Bajío, Leon, Guanajuato, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-2020-1001-155
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Acute Myocardial Infarction; Cardiovascular Morbidity; Heart Failure; Angina, Unstable
Keywords: Acute myocardial infarction; Dapagliflozin; mayor adverse cardiovascular events
MeSH Terms: conditions — Heart Failure; Angina, Unstable | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Asses the effect of Dapagliflozin on mayor adverse cardiovascular effects in patients with acute myocardial infarction compared against placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Dapagliflozin 10 mg every 24 hours for 12 months
  Interventions: Drug: Dapagliflozin 10Mg Tab
- Control Group (Placebo Comparator): 1 placebo tablet every 24 hours for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10Mg Tab — patients who meet the inclusion criteria will be randomized to receive dapagliflozin 10 mg every 24 hours for 12 months
  Arms: Intervention Group
Drug: Placebo — patients meeting the inclusion criteria will be randomized to receive a placebo solution every 24 hours for 12 months
  Arms: Control Group

SUMMARY:
The actual evidence is solid about the use of de SGLT2-inhibitors in wide spectrum of cardiorenal targets, which has been shown in a great amount of randomized clinical trials compared with placebo. At present it must be taken into account as first line treatment in patients with DM2, even their security profile has allowed the use in patients without diagnosis of DM2, since they have be shown a beneficial cardioprotect effects. Most studies support they use in patients with high cardiovascular risk, nevertheless, their use in patients with recent diagnosis of ischemic hearth disease its limited, being the latter entity the most frequent etiology found in patients who develop chronic hearth failure either as part of heart attack or unstable angina.

DETAILED DESCRIPTION:
According with the World Health Organization, cardiovascular disease is the leading cause of mortality in the world, estimating 17.9 millions of deaths a year. The cardiovascular disease are a group of disorders of the hearth and the blood vessels including coronary artery disease, cerebrovascular disease, rheumatic hearth disease and other conditions. Four out of five deaths attributed to cardiovascular cause are related to acute myocardial infarction and cerebrovascular disease and one third of this deaths occur in persons younger than 70 years.

The concept of acute coronary syndrome includes the ST elevation myocardial infarction who presents a ST elevation in two contiguous leads or complete left branch bundle block instead patients who presents without ST elevation in the electrocardiogram they are usually classified as Non ST elevation acute myocardial infarction.

The optimum treatment of the STEMI must be based in the utilization of networks between hospitals with different technology levels connected by an efficient y prioritized ambulance system. The objective of this networks is to provide an efficient medical attention, reduce the lag time and to get better the clinical results. The percutaneous coronary intervention is the preferred treatment of reperfusion for the patients with acute myocardial infarction on the first 12 hours after the development of symptoms, provided it can be done quickly (120 minutes since the diagnosis). In some circumstances, the PCI is not an option, then the fibrinolysis could be started immediately.

Most patients with ischemic heart disease are carriers of DM2. The DM2 is associated to an increase 3 times the risk of cardiovascular disease being this the principal cause of morbidity and mortality in this patients. Further, more than 40% of the patient with DM2 develops diabetic nephropathy and this increase strongly the risk of poor cardiovascular outcomes.

Improve the glycemic control in patients with DM2 has been a major objective in the clinical practice for decades, abreast to a reduction of the multifactorial cardiovascular risk. On randomized trials, controlled with placebo, the sodium-glucose linked transported inhibitors type 2 have shown convincingly improve the cardiovascular results, including a reduction in cardiovascular death and particularly, the reduction in the occurrence of heart failure leading to hospitalization . The consistent evidence of the beneficial cardiovascular effects of SGLT-2 inhibitors has led to recommend it in international papers for patients with DM2 and cardiovascular disease in addition to metformin, regardless of their basal levels of glycated hemoglobin.

The clinical trial EMPAREG OUTCOME in patients with DM2 and cardiovascular disease who receive a standard medical treatment shown a reduce in risk of MACE with empagliflozin compared with placebo, conferred mainly by a reduction in cardiovascular death. Mortality from all causes fell as well the risk of hospitalization associated to hearth failure. The CANVAS PROGRAM in patients with DM2 and high cardiovascular risk (66% had cardiovascular disease) shown also a reduction of risk of MACE with the use of canagiflozin compared against placebo, though the reduction on the risk of cardiovascular death and mortality by all causes didn't reach statistical significance.

The clinical trial DAPAHF included patients with LVEF of 45% and DM2 diagnosis. During the follow up (18.2 months) the patients aleatory assigned to receive dapagliflozin (in addition to standard medical therapy) had a significant reduction of 26% in risk of death from cardiovascular cause or deterioration of heart failure compared with placebo group, with a reduction of 18% of cardiovascular death. The amount of the effect were similar between patients with or without DM2, indicating a new beneficial mechanism that goes beyond glycemic control.

The SGLT-2 inhibitors effectively increase glycosuria, improve glycemic control and reduce the corporal mass index due to calorie loss. In addition, promote sodium excretion trough urine early (with a reduction in the plasmatic volume and increase in hematocrit), reduce the systemic blood pressure, and reduce the glomerular hyperfiltation and albuminuria. It is uncertain which of this mechanisms underlies the cardiovascular and renal benefits that had been shown in the big clinical trials but probably the sodium excretion trough urine early followed by a change in tisular sodium give a back up to protect against the decompensation against heart failure and the studies support this includes in patients without diagnosis of DM2. Other beneficial mechanisms includes a reduction in the inflammation mediated by adipose tissue and production of pro inflammatory cytokines, reduction in oxidative stress, inhibition of the exchanger Na+ / H+ of the myocardium and reduced levels of serum uric acid.

ELIGIBILITY:
Inclusion Criteria:

* Male and female IMSS eligible patients over 18 years of age
* Meet the criteria of the fourth definition of ST-segment elevation myocardial infarction
* Known with diabetes mellitus 2 or newly diagnosed diabetes according to ADA criteria

Exclusion Criteria:

* Patients diagnosed with Type 1 Diabetes Mellitus
* Patients on chronic replacement therapy for renal function through peritoneal dialysis or hemodialysis
* Patients who have recently undergone immunosuppressive therapy
* Patients with a history of recurrent urinary tract infection
* Patients known to be allergic to SGLT-2 inhibitors
* Patients presenting as sudden aborted death
* Patients who after percutaneous coronary intervention require orotracheal intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Mayor adverse cardiovascular effects | 12 months
  To assess the presence of myocardial infarction, stroke and death from cardiovascular causes in post-infarction patients during the study follow-up

SECONDARY OUTCOMES:
Left ventricular ejection fraction | 12 months
  Evaluate baseline left ventricular ejection fraction in post-infarct patients and 12 months of treatment
Chronic heart failure | 12 months
  Evaluate the effect of Dapagliflozin on the development of chronic heart failure that deserves hospitalization
Post infarction angina | 12 months
  Evaluate the effect of Dapagliflozin on the development of post infarction angina
Mortality due to cardiovascular cause | 12 months
  Assess the presence of mortality due to cardiovascular causes during the study follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Hilda E Macias Cervantes, Master in Clinical Research, Principal Investigator — Unidad Médica de Alta Especialidad No. 1 Bajío, Boulevard Adolfo López Mateos esquina Insurgentes S/N, colonia Los Paraísos, Leon, Guanajuato, Mexico, 37260; German R Bautista Lopez, Cardiology, Study Director — Unidad Médica de Alta Especialidad No. 1 Bajío, Boulevard Adolfo López Mateos esquina Insurgentes S/N, colonia Los Paraísos, Leon, Guanajuato, Mexico, 37260; Luis J Gonzalez, Cardiology Resident, Study Chair — Unidad Médica de Alta Especialidad No. 1 Bajío, Boulevard Adolfo López Mateos esquina Insurgentes S/N, colonia Los Paraísos, Leon, Guanajuato, Mexico, 37260; Rodolfo Guardado Mendoza, Endocrinologist, Study Director — Unidad de Investigación Metabólica, Universidad de Guanajuato, Boulevard Cañaveral 1001, fracciones de los Aguirre, CP 37672, León, Guanajuato, México; Gabriel Fernandez Yañez, Cardiology Resident, Study Chair — Unidad Médica de Alta Especialidad No. 1 Bajío, Boulevard Adolfo López Mateos esquina Insurgentes S/N, colonia Los Paraísos, Leon, Guanajuato, Mexico, 37260
Locations (1):
- Unidad Medica de Alta Especialidad No. 1, Bajío, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Alpert JS, Thygesen K, Antman E, Bassand JP. Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. J Am Coll Cardiol. 2000 Sep;36(3):959-69. doi: 10.1016/s0735-1097(00)00804-4. PMID 10987628
- [Result] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284
- [Result] Grupo de Trabajo de la Sociedad Europea de Cardiologia (ESC) sobre el manejo del infarto agudo de miocardio con elevacion del segmento ST (IAMCEST). Rev Esp Cardiol. 2009 Mar;62(3):293.e1-293.e47. doi: 10.1016/S0300-8932(09)70373-2. Epub 2009 Mar 19. No abstract available. English, Spanish. PMID 23040488
- [Result] Armstrong PW, Gershlick AH, Goldstein P, Wilcox R, Danays T, Lambert Y, Sulimov V, Rosell Ortiz F, Ostojic M, Welsh RC, Carvalho AC, Nanas J, Arntz HR, Halvorsen S, Huber K, Grajek S, Fresco C, Bluhmki E, Regelin A, Vandenberghe K, Bogaerts K, Van de Werf F; STREAM Investigative Team. Fibrinolysis or primary PCI in ST-segment elevation myocardial infarction. N Engl J Med. 2013 Apr 11;368(15):1379-87. doi: 10.1056/NEJMoa1301092. Epub 2013 Mar 10. PMID 23473396
- [Result] Cantor WJ, Fitchett D, Borgundvaag B, Ducas J, Heffernan M, Cohen EA, Morrison LJ, Langer A, Dzavik V, Mehta SR, Lazzam C, Schwartz B, Casanova A, Goodman SG; TRANSFER-AMI Trial Investigators. Routine early angioplasty after fibrinolysis for acute myocardial infarction. N Engl J Med. 2009 Jun 25;360(26):2705-18. doi: 10.1056/NEJMoa0808276. PMID 19553646
- [Result] Matheus AS, Tannus LR, Cobas RA, Palma CC, Negrato CA, Gomes MB. Impact of diabetes on cardiovascular disease: an update. Int J Hypertens. 2013;2013:653789. doi: 10.1155/2013/653789. Epub 2013 Mar 4. PMID 23533715
- [Result] Cowie MR, Fisher M. SGLT2 inhibitors: mechanisms of cardiovascular benefit beyond glycaemic control. Nat Rev Cardiol. 2020 Dec;17(12):761-772. doi: 10.1038/s41569-020-0406-8. Epub 2020 Jul 14. PMID 32665641
- [Result] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608
- [Result] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Result] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829